CLINICAL TRIAL: NCT02148094
Title: Closing a Critical HIV Prevention Gap: Demonstrating Safety and Effective Delivery of Daily Oral Pre-exposure Prophylaxis (PrEP) as Part of an HIV Combination Preventive Intervention for Sex Workers in Kolkata and Mysore-Mandya, India
Brief Title: Demonstrating Safety and Effective Delivery of Daily Oral Pre-exposure Prophylaxis (PrEP) for Sex Workers in India
Acronym: PrEP-India
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: World Health Organization (Other); DMSC (Unknown); Ashodaya Samithi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2014:050
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2016-10

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; India; Prevention; Female sex workers; PrEP; Pre-exposure prophylaxis; Truvada; Tenofovir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Truvada (Experimental): Participants will be initiated on PrEP and asked to select one of two PrEP delivery options. Participants will return to the study site every three months for an additional follow-up visit. At follow-up visits, participants will receive HIV testing and counselling, pregnancy testing, syndromic screening for STIs, and clinical diagnosis of adverse events. Those who test HIV-positive will be discontinued on PrEP, exited from the study and referred for HIV care and treatment. Those who have an adverse event will be clinically evaluated to determine whether they should suspend PrEP use and will be provided with the appropriate management for the adverse event. Participants who test HIV-negative will receive patient-centred counselling around PrEP.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — The demonstration project will use a prospective cohort design, enrolling individuals and following them up at multiple intervals over the course of 16 months. Study participants will be asked to take one tablet of Truvada daily, as HIV Pre-Exposure Prophylaxis, over this period. They will be asked to attend 7 regular visits at the project sites over the course of the project. In between visits, they will receive peer educator home visits every other day, as part of regular DMSC (Kolkata) and Ashodaya (Mysore/Mandya) outreach prevention activities. We plan to enroll 2000 female sex workers equally split between the two sites.
  Other Names: emtricitabine and tenofovir disoproxil fumarate

SUMMARY:
Female sex workers (FSWs) in India are at high risk of HIV infection, and while correct and consistent condom use is an effective means of preventing HIV transmission, many FSWs have difficulty insisting on their use. Alternative HIV prevention options are needed for FSWs who are unable to correctly and consistently use condoms with their clients or regular partners. Oral pre-exposure prophylaxis (PrEP) may be an important tool to fill this critical prevention gap, and a demonstration project is required to assess the impact and feasibility of the use of PrEP as an HIV prevention intervention among most at risk FSWs in India.

The proposed project will take place at two sites in India and will assess the use of a risk assessment tool to identify FSWs who would most benefit from PrEP, collect information about the reasons why FSWs choose to accept or decline PrEP, evaluate two different PrEP delivery strategies (weekly clinic pick-up or home delivery by peer educators every second day), monitor adherence to and discontinuation of PrEP, and evaluate unintended consequences of the use of PrEP in these communities (e.g. reduction of condom use, drug side effects or adverse events, social harms or resistance). To ensure the safety of study participants, a community advisory board will be set up and will meet regularly to inform study staff of any concerns that the community may have related to the study, so that the study staff can respond in a timely manner. A data safety and monitoring board will also be established to monitor participant safety.

DETAILED DESCRIPTION:
This PrEP demonstration study is designed to assess the feasibility and impact of delivering PrEP in addition to the existing package of HIV prevention interventions available to female sex workers in India. The study aims to: 1) identify female sex workers in need of HIV prevention and willing to take PrEP; 2) evaluate sustained uptake and adherence to oral PrEP; 3) assess safe delivery of PrEP; and 4) demonstrate effective delivery of PrEP within the context of the National Program of Targeted Interventions. The study will be implemented in two regions and among two typologies of female sex workers in India: brothel-based FSWs in Kolkata and FSWs operating from different settings in Mysore and Mandya.

Outcome 1: Identification of female sex workers in need of HIV prevention and willing to take oral PrEP For optimal delivery with limited resources, it is critical to provide HIV prevention strategies such as PrEP to populations at greatest risk of infection. Female sex workers are an important population for HIV prevention in India, prioritized as a "core high risk group" for targeted interventions by the India National AIDS Control Organization (NACO) (NACO 2013 annual report). In particular, some FSWs report inconsistent condom use and have unmet needs for HIV prevention (Ramesh, 2010; Reza-Paul, 2008). For example, these women may be less empowered or able to consistently demand condom use by their clients or may wish to become pregnant. PrEP has the potential to be an additional, more acceptable and effective HIV prevention method for female sex workers who have difficulty using condoms consistently.

This study proposes the development and use of a risk screening tool to identify female sex workers who are most vulnerable to HIV. This tool will guide recruitment into the demonstration study and could later assist health providers in deciding who will benefit most from PrEP for HIV prevention. In addition, this study will assess the proportion of FSWs identified by the risk screening tool who are willing to take PrEP. Quantitative and qualitative evaluations will identify factors related to the decision to initiate PrEP as well as reasons why FSWs decline PrEP.

Outcome 2: Sustained uptake and adherence to oral PrEP among female sex workers Similar to all medications, sustained uptake and adherence to PrEP is fundamental for efficacy in preventing HIV acquisition. In the four clinical trials of oral PrEP that demonstrated efficacy, study participants with high adherence had the greatest protection from HIV (Baeten 2012, Choopanya 2013, Grant 2010, Thigpen 2012). Likewise, across PrEP trials, there was a clear relationship between higher efficacy and a greater proportion of participants with study drug detectable in their blood. Two randomized clinical trials of daily oral PrEP among heterosexual women in Africa found no efficacy for HIV prevention; poor adherence to PrEP most likely explains these results (Marrazzo 2013, Van Damme 2012). For example, drug level testing in the FEM-PrEP Study found that less than 40% of a random sample of HIV negative women in the PrEP arm of the study had detectable levels of PrEP in their blood (Van Damme 2012). Analyses of high-risk subgroups of study participants in the Partners PrEP Study found PrEP efficacy estimates ranged from 64 to 84%, showing consistently high efficacy of PrEP in preventing HIV across various higher risk groups, including women (Murnane 2013).

Preliminary community awareness campaigns for PrEP among female sex workers in Kolkata found high interest in PrEP - approximately 80% reported willingness to take daily, oral PrEP. Sex workers in Mysore-Mandya are engaged in series of consultations where information related to PrEP as a tool for combination prevention is being discussed and questions or concerns related to PrEP addressed. In both places, initial observations show that there are some sex workers (e.g. those who are on long time contracts, those with overnight clients where sometimes the number of clients are not disclosed, those who want to be pregnant, and those who do not use condoms with their regular partners) expressed interest in being part of the demonstration project.

This PrEP demonstration study will assess the acceptability and feasibility of two approaches to PrEP delivery: 1) peer educator delivery every other day; or 2) weekly clinic pick-up. Study staff will measure PrEP initiation, adherence and discontinuation. They will record these events in participant records, and quarterly visits will be used to assess adherence through biological tests and questionnaires. PrEP will be delivered as part of a package of HIV prevention services, and therefore use of other prevention strategies, such as condom use, will also be monitored. The full package of prevention services will continue to be provided to FSWs with the support of India's national government and in accordance with national guidelines.

Data on drug adherence and condom use will be collected through various means. An ethnographic study will be designed to understand factors that may promote or impede adherence to PrEP, as well as changes in risk behaviour (reduction in condom use). In addition to this, peer educators will use a pictorial tool to document these items (e.g., frequency and patterns of sexual activity, condom use, and PrEP use). The study will also include a biological measure of PrEP adherence through the assessment of drug-levels in the blood.

Regular counselling about HIV prevention and PrEP will be provided to study participants to promote adherence. In a sub-sample of study participants, an electronic adherence monitoring device to measure and promote adherence, Helping Hands, will be tested (De Blaser 2010). The Helping Hands device is complimented by a web platform that illustrates patient-specific data to monitor dosing history and adherence patterns.

Outcome 3: Oral HIV PrEP as part of a combined prevention package delivered safely for female sex workers Four randomized controlled trials have demonstrated that daily, oral PrEP is safe for HIV-uninfected women in a wide range of settings; these antiretrovirals have been proven safe for HIV-infected women for many years of use. The most common side effects of FTC/TDF are minor and short-lived (i.e. first several weeks). This study will provide evidence for the safe delivery of oral PrEP to female sex workers in brothel and street-based settings in India. Quarterly clinic visits will assess physical health, side effects, adverse events and any other social harms or concerns with PrEP use. This study will invest in continuous engagement with communities of female sex workers according to good participatory practice guidelines to provide correct information about PrEP, keep communities continuously engaged, and maintain adherence to PrEP.

A community advisory board (CAB) and a Data Safety and Monitoring Board (DSMB) will be set up. The CAB will meet monthly and on an as needed basis. It will inform study staff of any concerns that the community may have related to the study, so that the study staff can respond in a timely manner. The CAB members will be close to the community and will be able to respond to community concerns by calling meetings to address issues in a timely manner. The DSMB will be set up to ensure that the rights of the study participants are safeguarded in a transparent fashion, and to monitor their safety by scrutinizing any adverse events. The DSMB will also help to respond to concerns raised by the CAB. The DSMB will include an ethicist, a human rights lawyer, representatives from University of Manitoba, WHO and UNAIDS, representatives from the global network of sex workers, and a statistician. In addition, ongoing qualitative research and monitoring by research staff, as well as outreach by peer educators, will attempt to identify any community resistance, rumours or actual harms, and respond in an appropriate manner.

Outcome 4: Effective delivery of oral HIV PrEP demonstrated in context of National Program of Targeted Interventions This study proposes to deliver PrEP within the context of the National Program of Targeted Interventions in order to demonstrate that PrEP is feasible in "real world" settings. DMSC and Ashodaya currently implement targeted intervention programs for female sex workers in Kolkata and Mysore/Mandya, respectively. These programs provide outreach by peer educators and outreach workers, clinic services (e.g. HIV testing and counseling, STI screening and treatment), and referrals for HIV care and treatment for brothel- and street-based FSWs. This study will evaluate the addition of PrEP to this existing service delivery model. It will also show willingness of participants to enroll in a demonstration study and to use oral PrEP without reimbursements or incentives for participation.

Study findings can inform national and local government's decision to adopt PrEP as a new HIV prevention strategy. Development of HIV prevention packages, provider training, quality management and service delivery guidelines in line with national systems will provide guidance for real life implementation of PrEP, and also contribute to the larger goal of providing standards for the delivery of HIV prevention interventions.

Risk Mitigation Identification of willing participants: The development of a tool to correctly identify those FSWs at continued risk of HIV infection does not ensure that those women will be willing to take PrEP. Though initial interest in PrEP is strong in Sonagachi among FSWs in general, women at highest risk may be different. A feasibility study to identify levels of awareness about PrEP, perceptions and misconceptions about PrEP, and optimum ways to present PrEP accurately to identify those women at greatest need with greatest interest in using PrEP is about to begin in Mysore.

Research ethics: All study materials will be submitted for approval by the institutional review boards of Durbar Mahila Samanwaya Committee (DMSC) Ethical Committee, the World Health Organization (WHO) Ethics Review Committee (ERC), the University of Manitoba (UM) Health Research Ethics Board (HREB), and by the Indian Council on Medical Research (ICMR) through the Health Ministry's Screening Committee (HMSC). The procedures, risks, and benefits of study participation will be explained to all potential study participants and informed consent will be obtained from those who are willing to participate prior to their participation in the study. The project will follow all guidelines for human subjects research as mandated by the Government of India, as this is the location of the proposed project. In addition to this, a Data Safety and Monitoring Board will be established at Ashodaya to monitor the safety of participants and the scientific integrity of the study across all study sites.

Community advisory board (CAB): A community advisory board will be set up in each study site, and will meet regularly to inform study staff and the DSMB of any concerns that the community may have related to the study, so that the study staff can respond in a timely manner.

Data Safety and Monitoring Board (DSMB): A DSMB will be established to ensure that the rights of all study participants from each site, Ashodaya and DMSC, are safeguarded, and to monitor their safety by scrutinizing any adverse events. They will also respond to concerns raised by the CABs from each site. The DSMB will include an ethicist, a human rights lawyer, representatives from the University of Manitoba, WHO and UNAIDS, representatives from the global network of sex workers, and a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as a current FSW
* Age 18 and older
* Self-reported interest in and willingness to take PrEP
* Score cutoff on risk screening tool / PrEP indication tool
* HIV-negative test at time of enrollment (per testing algorithm)
* No clinical signs of acute HIV infection
* Hepatitis-B virus antigen negative (upon screening)
* Creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula) (upon screening)
* Not currently taking PrEP or enrolled in another PrEP demonstration project
* Negative urine pregnancy test at time of enrollment
* Lives within the catchment area of the project site and no plans to move away from the project area in the next 16 months

Exclusion Criteria:

* Under 18
* Does not meet inclusion criteria

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1325 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Sustained uptake and adherence to oral PrEP among female sex workers | 24 months
  We will assess the acceptability and feasibility of two approaches to PrEP delivery: 1) peer educator delivery every other day; or 2) weekly clinic pick-up. Study staff will measure PrEP initiation, adherence and discontinuation. They will record these events in participant records, and quarterly visits will be used to assess adherence through biological tests and questionnaires. PrEP will be delivered as part of a package of HIV prevention services, and therefore use of other prevention strategies, such as condom use, will also be monitored. Data on drug adherence and condom use will be collected through various means. An ethnographic study will be designed to understand factors that may promote or impede adherence to PrEP, as well as changes in risk behaviour (reduction in condom use). In addition to this, peer educators will use a pictorial tool to document these items (e.g., frequency and patterns of sexual activity, condom use, and PrEP use).

SECONDARY OUTCOMES:
Identification of female sex workers willing to take PrEP | 18 months after study commencement
  We propose to develop and use of a risk screening tool to identify female sex workers who are most vulnerable to HIV. This tool will guide recruitment into the demonstration study and could later assist health providers in deciding who will benefit most from PrEP for HIV prevention. In addition, this study will assess the proportion of FSWs identified by the risk screening tool who are willing to take PrEP. Quantitative and qualitative evaluations will identify factors related to the decision to initiate PrEP as well as reasons why FSWs decline PrEP
Oral HIV PrEP as part of a combined prevention package delivered safely for female sex workers | 24 months
  The most common side effects of FTC/TDF are minor and short-lived (i.e. first several weeks). Quarterly clinic visits will assess physical health, side effects, adverse events and any other social harms or concerns with PrEP use. This study will invest in continuous engagement with communities of female sex workers according to good participatory practice guidelines to provide correct information about PrEP, keep communities continuously engaged, and maintain adherence to PrEP. A community advisory board (CAB) and a Data Safety and Monitoring Board (DSMB) will be set up. The CAB will meet monthly and on an as needed basis. The DSMB will be set up to ensure that the rights of the study participants are safeguarded in a transparent fashion, and to monitor their safety by scrutinizing any adverse events.
Effective delivery of oral HIV PrEP demonstrated in context of National Targeted Interventions | 24 months
  This study proposes to deliver PrEP within the context of the National Program of Targeted Interventions in order to demonstrate that PrEP is feasible in "real world" settings. DMSC and Ashodaya currently implement targeted intervention programs for female sex workers in Kolkata and Mysore/Mandya, respectively. These programs provide outreach by peer educators and outreach workers, clinic services (e.g. HIV testing and counseling, STI screening and treatment), and referrals for HIV care and treatment for brothel- and street-based FSWs. This study will evaluate the addition of PrEP to this existing service delivery model. It will also show willingness of participants to enroll in a demonstration study and to use oral PrEP without reimbursements or incentives for participation.

CONTACTS AND LOCATIONS:
Overall Officials: Sushena Reza-Paul, MBBS, Principal Investigator — University of Manitoba, Ashodaya Samithi; Smarajit Jana, MBBS, Principal Investigator — DMSC
Locations (2):
- India (2):
  - Ashodaya Samithi clinic, Mysore, Karnataka
  - DMSC Clinic, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No